CLINICAL TRIAL: NCT06972017
Title: Peri-Operative Surgical Care Optimisation for Patients Requiring Emergency Surgery
Acronym: PERI-SCOPES
Status: Not yet recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Bowel Research UK (Unknown); NHS Lothian (Other Government); NHS Grampian (Other Government); NHS Tayside (Other Government); University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: UGN23SG190; PhD_23017 (Other Grant/Funding Number: Bowel Research UK)
Record Dates: First submitted 2025-04-17; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Quality of Life (QOL); Decision Making; Emergency General Surgery
Keywords: Quality of Life; Decision-making; NoLap; EmLap; Emergency General Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- EmLap patients: Patients who have underwent Emergency General Surgery
- NoLap patients: Patients who have needed but not undergone Emergency General Surgery.
- Families/Supporters: Family or supporter nominated by the patient participant to participate in the study alongside them.
- Consultants: Consultants who actively participate in Emergency General Surgery in a UK-based Hospital (Surgeons, Anaesthetists, Intensivists)

SUMMARY:
Emergency General Surgery (EGS) is an umbrella term which describes all patients presenting to hospital with an acute abdominal problem. Patients can have various conditions requiring emergency operations. EGS is one of the most common reasons for an emergency admission in the UK.

EGS is often referred to as "high-risk" surgery. For those patients who do survive after their surgery, many struggle with frailty and new medical problems resulting in a reduction in their quality of life (QoL).

The goal of this observational study is to explore QoL and decision-making in EGS through questionnaires and interviews with patients, families/supporters and consultants working in EGS.

Workstream 1 will involve patients and families/supporters. Workstream 2 will involve consultants.

The investigators are interested in patients who have either undergone EGS (EmLaps) or have needed but not undergone EGS (NoLaps). The investigators are interested in exploring participants (patients, families/supporters and consultants) experiences of this EmLap vs NoLap decision.

The main questions the investigators want to answer are:

* What is the long-term QOL of EmLap/NoLap patients and their family/supporters?
* How do patients and their family/supporters describe their experience of decision-making in EGS?
* What are consultant's experiences and views on decision-making in EGS?

Workstream 1 participants (patients and family members/supporters) will complete questionnaires and take part in interviews at different time-points following their decision (1 month/3 months/ 9-12 months). Questionnaires and interviews will explore QoL and decision-making in EGS.

Consultant participants will be asked to complete an online survey and/or take part in an individual interview. Both will explore decision-making in EGS.

ELIGIBILITY:
Group 1 and 2: EmLap and NoLap patients (up to 30 participants)

Patient inclusion/exclusion criteria should mirror NELA inclusion/exclusion criteria and NELA NoLap guidelines. NELA is the "National Emergency Laparotomy Audit" which recruits patients in Wales and England and there inclusion/exclusion criteria are widely accepted for use in Emergency General Surgery research.

Inclusion criteria

* Age >65 years old
* Able to communicate in English
* Cognitively able to complete the survey/interviews
* Able to provide informed, voluntary consent
* First line treatment is expedited, urgent or emergency abdominal surgery on the gastrointestinal tract
* Surgery can be laparoscopic or open approach

Exclusion criteria

* Age <65 years old
* NoLaps should be excluded if management involved interventional radiology or endoscopic procedures
* Patients who are offered a period of conservative treatment are not automatically NoLap if surgery may ultimately be offered
* Diagnosis of dementia or long-standing cognitive impairment
* Elective laparotomy/laparoscopy
* Diagnostic laparotomy/laparoscopy where no subsequent procedure is performed (however, if no procedure is performed because of inoperable pathology, then include)
* All surgery involving the appendix or gallbladder, including any surgery relating to complications
* Non-elective hernia repair without bowel resection or division of adhesions
* Non-elective formation of colostomy or ileostomy
* Trauma surgery (blunt or penetrating), vascular surgery, obstetric/gynaecological surgery or transplant surgery
* Surgery for pathology of oesophagus, spleen, renal tract, kidneys, liver, gallbladder and biliary tree, pancreas or urinary tract

Group 3: Families/Supporters (up to 30 participants) Inclusion criteria

* Identified by the patient participant (only approached if nominated by patient)
* Age >18 years old
* Able to communicate in English
* Cognitively able to complete the survey/interviews
* Able to provide informed, voluntary consent

Exclusion criteria

* Age<18 years old
* Lack of patient consent to family/supporter involvement

Group 3: Consultants (interview:12-20 participants/survey: minimum 52 participants) Inclusion criteria

* Key decision-makers will be identified in workstream 1 (likely: surgeons, intensivists and anaesthetists)
* Post-CCT (Certificate of Completion of Training)
* Participate in active on-call for EGS in a UK-based Hospital where they make decisions in EGS regularly

Exclusion criteria

• Consultants not done >2 years of on-call

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Project will recruit EmLap and NoLap patients from the 6 sites across Scotland with the highest EmLaps per year (Queen Elizabeth University Hospital, Glasgow Royal Infirmary, Royal Alexandra Hospital, Aberdeen Royal Infirmary, Ninewells Hospital, Edinburgh Royal Infirmary).
  Consultants will be recruited from UK only.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL) | 1 year
  The primary aim of workstream 1 is to report on the long-term QoL of EmLap and NoLap patients and their families/supporters. For this, participants will complete validated QoL questionnaires within 4 weeks of EmLap/NoLap decision then again at 3 and 9-12 months post-decision.
  Questionnaires will include European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) which will specifically quantify QoL. Maximum score= 1. Minimum scores in the UK have been reported at -0.28. A higher score reflects a higher QoL.
Decision-making | 1 year
  The primary aim of workstream 2 is to describe and explore consultant experiences of decision-making in EGS through online survey and semi-structured interviews.

SECONDARY OUTCOMES:
Decision-making | 1 year
  Semi-structured interviews with patients and families/supporters will allow us to explore their experience and views of decision-making in EGS.
Consultant specialities involved in decision-making | 1 year
  Workstream 1 will clarify which specialties are involved in the EGS decision-making process to allow recruitment for workstream 2.
  We will specifically clarify the number of EGS decisions which involve
  * consultant surgeon
  * consultant anaesthetist
  * consultant intestivist
Patient Reported Outcome Measurements (PROMs) for Emergency General Surgery | 1 year
  The results from workstream 1 will inform the development of PROMs for EGS. These PROMS will include a number of specific EGS related questions developed from our study results.
Patient Reported Experience Measurements (PREMs) for Emergency General Surgery | 1 year
  The results from workstream 1 will inform the development of PREMs for EGS. These PREMS will include a number of specific EGS related questions developed from our study results.

IPD SHARING:
Plan to Share IPD: No
Psuedonymized personal data will retained only for as long as required for processing (1 year after project has ended). Only depersonalised anonymous research data will be stored for a longer period of time and shared with other researchers.